CLINICAL TRIAL: NCT00717418
Title: Efficacy Study of Cyclosporine Ophthalmic Emulsion in Patients With Dry Eye Disease
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: R.E.S.T.O.R.E.
Record Dates: First submitted 2008-07-14; First posted 2008-07-17 (Estimated); Results first posted 2012-01-12 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2011-12

CONDITIONS: Keratoconjunctivitis Sicca
MeSH Terms: conditions — Keratoconjunctivitis Sicca | interventions — Cyclosporins; Lubricant Eye Drops

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: * cyclosporine ophthalmic emulsion 0.05%
  * artificial tears
  Interventions: Drug: cyclosporine ophthalmic emulsion 0.05%, artificial tears

INTERVENTIONS:
Drug: cyclosporine ophthalmic emulsion 0.05%, artificial tears — one drop, twice a day in each eye
  Other Names: Restasis®

SUMMARY:
This study will evaluate the efficacy of cyclosporine ophthalmic solution vs. other non-prescription treatments in patients with dry eye disease. Patient and physician assessments completed at baseline, at each follow-up visit (follow-up visits are variable as per physician discretion) and at final follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dry eye disease
* Currently using artificial tears daily
* Male or female of legal age of consent
* Normal lid position and closure

Exclusion Criteria

* Patients currently using cyclosporine ophthalmic emulsion 0.05%
* Participation in other investigational drug or device study
* Any current or previous topical ophthalmic or oral cyclosporine use within the last three years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients can either:
  1. be newly diagnosed or changing therapies and require, in the judgment of the treating physician, a prescription treatment
  2. have insufficiently controlled dry eye symptoms necessitating use of over-the-counter treatments
Sampling Method: Non-Probability Sample
Enrollment: 781 (Actual)
Dates: Start 2004-09; Primary Completion 2006-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Wilson, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Treatment for this study was per normal clinical practice and not assigned.
Groups:
- Restasis® Alone: cyclosporine ophthalmic emulsion 0.05%
Period: Baseline
Arm/Group | Restasis® Alone | Artificial Tears Alone | Combination Treatments | Missing Treatment Information
Started | 180 | 74 | 508 | 19
Completed | 180 | 74 | 508 | 4
Not Completed | 0 | 0 | 0 | 15
Period: 1-Year Follow-Up
Arm/Group | Restasis® Alone | Artificial Tears Alone | Combination Treatments | Missing Treatment Information
Started | 180 | 74 | 508 | 4
Completed | 33 | 23 | 74 | 0
Not Completed | 147 | 51 | 434 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Restasis® Alone | Artificial Tears Alone | Combination Treatments | Missing Treatment Information | Total
Number analyzed (Participants) | 180 | 74 | 508 | 19 | 781
Age Continuous [Median (Full Range); unit: years] | 55.0 [19 to 91] | 64.5 [28 to 87] | 60.0 [18 to 96] | 61.0 [26 to 87] | 60.0 [18 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 62 | 425 | 15 | 627
  Male | 55 | 12 | 83 | 4 | 154

OUTCOME MEASURES:

1. Primary Outcome: Ocular Surface Disease Index (OSDI) Total Score at Baseline
Description: The OSDI consists of 12 questions to assess visual function, ocular symptoms and environmental triggers related to dry eye. Each of the 12 questions is assessed using a 5-point scale (0=none of the time; 4 = all of the time) which is converted to a total score between 0-100. OSDI total scores of 0-12=normal (best), 13-22= mild ocular surface disease, 23-32 =moderate ocular surface disease, and 33-100=severe ocular surface disease (worst).
Time Frame: Baseline
Population: Intent-to-treat, which included all patients who started the study (completed baseline visit) and were assessed for this outcome measure. 16 subjects did not complete this outcome measure assessment and were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | All Patients
Number analyzed (Participants) | 750
Scores on a Scale | 40.3 (22.0)

2. Other Pre Specified Outcome: Schirmer's Test With and Without Anesthesia at Baseline
Description: Schirmer's Test with and without anesthesia at baseline. The Schirmer's test is performed on each eye with and without anesthesia (numbing eye drop). The amount of wetting produced by the eye was measured in millimeters using a graduated paper scale. The results indicate the presence of dry eye (Normal = greater than or equal to 15 millimeters (mm), Dry eye = less than 15 mm). A larger number correlates to better tear production, a smaller number correlates to reduced tear production.
Time Frame: Baseline
Population: Intent-to-treat, which included all patients who started the study (completed baseline visit).
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | All Patients
Number analyzed (Participants) | 766
millimeters (mm)
  Schirmer's Test with Anesthesia | 8.1 (6.3)
  Schirmer's Test without Anesthesia | 9.6 (7.9)

ADVERSE EVENTS:
Description: Serious adverse events and adverse events were not collected/assessed.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Due to actual dry eye treatment used, data were not interpretable by separate treatment arms. Hence, Outcomes are only reported as a single group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo